CLINICAL TRIAL: NCT03151811
Title: A Randomized, Controlled, Open-label, Phase 3 Study of Melflufen/Dexamethasone Compared With Pomalidomide/Dexamethasone for Patients With Relapsed Refractory Multiple Myeloma Who Are Refractory to Lenalidomide
Brief Title: A Study of Melphalan Flufenamide (Melflufen)-Dex or Pomalidomide-dex for RRMM Patients Refractory to Lenalidomide
Acronym: OCEAN
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor assessed all endpoints and collected Overall Survival data for another two years following the primary completion date of 03Feb2021.
Sponsor: Oncopeptides AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OP-103
Record Dates: First submitted 2017-05-09; First posted 2017-05-12 (Actual); Results first posted 2022-07-27 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2023-12

CONDITIONS: Multiple Myeloma
Keywords: Refractory Multiple Myeloma; Relapsed Multiple Myeloma; Melphalan flufenamide (Melflufen); Pomalidomide; Dexamethasone
MeSH Terms: conditions — Multiple Myeloma | interventions — melflufen; L-melphalanyl-p-L-fluorophenylalanine ethyl ester; pomalidomide; Dexamethasone; dexamethasone acetate; Calcium Dobesilate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Melflufen+Dexamethasone (Experimental): Melflufen 40 mg i.v. on Day 1 and dexamethasone 40 mg (20 mg for patients ≥ 75 years of age) on Days 1, 8, 15 and 22 of each 28-day cycle. Patients were to be treated until confirmed progression, unacceptable toxicity, or the patient or investigator decided it was not in the patient's best interest to continue.
  Interventions: Drug: Melflufen; Drug: Dexamethasone
- Arm B: Pomalidomide+Dexamethasone (Active Comparator): Pomalidomide 4 mg orally daily on Days 1 to 21 and dexamethasone 40 mg (20 mg for patients ≥ 75 years of age) on Days 1, 8, 15 and 22 of each 28-day cycle. Patients were to be treated until confirmed progression, unacceptable toxicity, or the patient or investigator decided it was not in the patient's best interest to continue.
  Interventions: Drug: Pomalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Melflufen — Intravenous infusion
  Other Names: Melphalan Flufenamide; Pepaxti
  Arms: Arm A: Melflufen+Dexamethasone
Drug: Pomalidomide — Oral capsules
  Other Names: Pomalyst; Imnovid
  Arms: Arm B: Pomalidomide+Dexamethasone
Drug: Dexamethasone — Oral tablets
  Other Names: Dex; Fortecortin; Decadron

SUMMARY:
This was a randomized, controlled, open-label, Phase 3 multicenter study which enrolled patients with RRMM following 2-4 lines of prior therapy and who were refractory to lenalidomide in the last line of therapy as demonstrated by disease progression on or within 60 days of completion of the last dose of lenalidomide. Patients received either melflufen+dex or pomalidomide+dex.

DETAILED DESCRIPTION:
This was a randomized, controlled, open-label, Phase 3 multicenter study which enrolled patients with RRMM following 2-4 lines of prior therapy and who were refractory to lenalidomide in the last line of therapy as demonstrated by disease progression on or within 60 days of completion of the last dose of lenalidomide.

Patients were randomized to either one of two arms:

Arm A: Melphalan flufenamide (Melflufen) 40 mg on Day 1 and dexamethasone 40 mg on Days 1, 8, 15 and 22 of each 28-day cycle.

Arm B: Pomalidomide 4 mg daily on Days 1 to 21 and dexamethasone 40 mg on Days 1, 8, 15 and 22 of each 28-day cycle.

Patients ≥ 75 years of age received a reduced dose of dexamethasone of 20 mg on Days 1, 8, 15 and 22 for both Arm A and Arm B.

Patients were to receive treatment until such time as there was documented disease progression, unacceptable toxicity, or the patient/treating physician determined it was not in the patient's best interest to continue.

Dose modifications and delays in therapy may have been implemented based on patient tolerability as detailed in the protocol. In the event of a cycle delay, unrelated to dexamethasone toxicity, it was recommended to continue dexamethasone weekly.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age 18 years or older
2. A prior diagnosis of multiple myeloma with documented disease progression requiring further treatment at time of screening
3. Measurable disease defined as any of the following:

   * Serum monoclonal protein ≥ 0.5 g/dL by protein electrophoresis.
   * ≥ 200 mg/24 hours of monoclonal protein in the urine on 24-hour electrophoresis
   * Serum free light chain ≥ 10 mg/dL AND abnormal serum kappa to lambda free light chain ratio
4. Received 2-4 prior lines of therapy, including lenalidomide and a PI, either sequential or in the same line, and is refractory (relapsed and refractory or refractory) to both the last line of therapy and to lenalidomide (≥ 10 mg) administered within 18 months prior to randomization. Refractory to lenalidomide is defined as progression while on lenalidomide therapy or within 60 days of last dose, following at least 2 cycles of lenalidomide with at least 14 doses of lenalidomide per cycle.
5. Life expectancy of ≥ 6 months
6. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
7. Females of child bearing potential (FCBP) must have a negative serum or urine pregnancy test prior to start of treatment. Participants must agree to ongoing pregnancy testing. All patients must be willing to comply with all requirements of the USA pomalidomide Risk Evaluation and Mitigation Strategy (REMS) program or the pomalidomide Pregnancy Prevention Plan (PPP).
8. Ability to understand the purpose and risks of the study and provide signed and dated informed consent.
9. 12-lead Electrocardiogram (ECG) with QT interval calculated by Fridericia Formula (QTcF) interval of ≤ 470 msec Fridericia Formula.
10. The following laboratory results must be met during screening and also immediately before study drug administration on Cycle 1 Day 1:

    * Absolute neutrophil count (ANC) ≥ 1,000 cells/mm^3 (1.0 x 10^9/L)
    * Platelet count ≥ 75,000 cells/mm^3 (75 x 10^9/L)
    * Hemoglobin ≥ 8.0 g/dl
    * Total Bilirubin ≤ 1.5 x upper limit of normal (ULN), or patients diagnosed with Gilberts syndrome, that have been reviewed and approved by the medical monitor.
    * Aspartate transaminase (AST /SGOT) and alanine transaminase (ALT/SGPT) ≤ 3.0 x ULN.
    * Renal function: Estimated creatinine clearance by Cockcroft-Gault formula ≥ 45 mL/min.
11. Must be able to take antithrombotic prophylaxis.
12. Must have, or be willing to have an acceptable central catheter. (Port a cath, peripherally inserted central catheter [PICC-line], or central venous catheter) (Insertion only required if randomized to Arm A).

Exclusion Criteria:

1. Primary refractory disease (i.e. never responded (≥ MR) to any prior therapy)
2. Evidence of mucosal or internal bleeding or platelet transfusion refractory
3. Any medical conditions that, in the Investigator's opinion, would impose excessive risk to the patient or would adversely affect his/her participating in this study.
4. Prior exposure to pomalidomide
5. Known intolerance to IMiDs.
6. Known active infection requiring parenteral or oral anti-infective treatment within 14 days of randomization.
7. Other malignancy diagnosed or requiring treatment within the past 3 years with the exception of adequately treated basal cell carcinoma, squamous cell skin cancer, carcinoma in-situ of the cervix or breast or very low and low risk prostate cancer in active surveillance.
8. Pregnant or breast-feeding females
9. Serious psychiatric illness, active alcoholism, or drug addiction that may hinder or confuse compliance or follow-up evaluation
10. Known human immunodeficiency virus or active hepatitis C viral infection
11. Active hepatitis B viral infection (defined as HBsAg+).

    * Patients with prior hepatitis B vaccine are permitted (defined as HBsAg-, Anti-HBs+, Anti-HBc-).
    * Non-active hepatitis B (HBsAg-, Anti-HBs+, Anti-HBc+) may be enrolled at the discretion of the investigator after consideration of risk of reactivation.
12. Concurrent symptomatic amyloidosis or plasma cell leukemia
13. POEMS syndrome
14. Previous cytotoxic therapies, including cytotoxic investigational agents, for multiple myeloma within 3 weeks (6 weeks for nitrosoureas) prior to randomization. IMiDs, PIs and or corticosteroids within 2 weeks prior to randomization. Other investigational therapies and monoclonal antibodies within 4 weeks of randomization. Prednisone up to but no more than 10 mg orally q.d. or its equivalent for symptom management of comorbid conditions is permitted but dose should be stable for at least 7 days prior to randomization
15. Residual side effects to previous therapy > grade 1 prior to randomization (Alopecia any grade and/or neuropathy grade 2 without pain are permitted)
16. Prior peripheral stem cell transplant within 12 weeks of randomization
17. Prior allogeneic stem cell transplantation with active graft-versus-host-disease.
18. Prior major surgical procedure or radiation therapy within 4 weeks of the randomization
19. Known intolerance to steroid therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 495 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2021-02-03 (Actual); Study Completion 2023-02-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pieter Sonneveld, Prof., Principal Investigator — Erasmus Medical Center
Locations (105):
- United States (14):
  - US17, Tucson, Arizona
  - US01, Fresno, California
  - US11, Gainesville, Florida
  - US12, Orange City, Florida
  - US-19, Plantation, Florida
  - US16, Boise, Idaho
  - US-24, Louisville, Kentucky
  - US13, Boston, Massachusetts
  - US-27, Hattiesburg, Mississippi
  - US-21, Salisbury, North Carolina
  - US-30, Winston-Salem, North Carolina
  - US06, Philadelphia, Pennsylvania
  - US15, Fort Sam Houston, Texas
  - US-18, Temple, Texas
- Austria (2):
  - AT-02, Linz
  - AT-01, Vienna
- Belgium (3):
  - BE-05, Edegem
  - BE-03, Liège
  - BE-02, Roeselare
- Czechia (5):
  - CZ-05, Brno
  - CZ-03, Hradec Králové
  - CZ-04, Olomouc
  - CZ-01, Ostrava
  - Cz-02, Cz-06, Prague
- DK01, Vejle, Denmark
- Estonia (2):
  - EE-01, Tallinn
  - EE-02, Tartu
- France (10):
  - FR04, Brest
  - FR-11, Cholet
  - FR01, Le Mans
  - FR05, Limoges
  - FR-07, Lyon
  - FR06, Lyon
  - FR03, Mulhouse
  - FR-09, Nice
  - FR-10, Périgueux
  - FR-08, Poitiers
- Greece (3):
  - Gr02, Gr03, Athens
  - GR04, Pátrai
  - GR01, Thessaloniki
- Hungary (4):
  - Hu02, Hu03, Hu04, Budapest
  - HU01, Debrecen
  - HU-06, Kaposvár
  - HU-05, Pécs
- Israel (6):
  - IL03, Jerusalem
  - IL01, Nahariya
  - IL05, Rehovot
  - IL02, Safed
  - IL04, Tel Aviv
  - IL06, Tel Aviv
- Italy (8):
  - IT07, Bergamo
  - IT02, Bologna
  - IT08, Brescia
  - It03, It09, Milan
  - IT06, Modena
  - IT04, Piacenza
  - IT05, Terni
  - IT01, Torino
- Lithuania (2):
  - LT-02, Kaunas
  - LT-01, Vilnius
- NL01, Rotterdam, Netherlands
- Norway (2):
  - NO-02, Ålesund
  - NO01, Oslo
- Poland (8):
  - PL03, Bialystok
  - PL02, Chorzów
  - PL06, Lodz
  - PL05, Lublin
  - PL-08, Olsztyn
  - PL07, Poznan
  - PL04, Rzeszów
  - PL-09, Torun
- Romania (2):
  - RO-02, Brasov
  - RO-01, Bucharest
- Russia (10):
  - RU-04, Izhevsk
  - Ru-11, Ru-14, Krasnoyarsk
  - RU-03, Moscow
  - RU-09, Nizhny Novgorod
  - RU-10, Novosibirsk
  - RU-06, Petrozavodsk
  - Ru-01, Ru-02, Ru-08, Ru-12, Ru-14, Saint Petersburg
  - RU-07, Samara
  - RU-13, Syktyvkar
  - RU-05, Yekaterinburg
- South Korea (4):
  - KR-06, Busan
  - KR-05, Daegu
  - KR-04, Hwasun
  - Kr-01, Kr-02, Kr-03, Seoul
- Spain (9):
  - ES11, Badalona
  - Es02, Es13, Es14, Barcelona
  - Es01, Es04, Es09, Madrid
  - ES-15, Málaga
  - Es07, Es12, Pamplona
  - ES10, Salamanca
  - ES03, Santa Cruz de Tenerife
  - ES08, Seville
  - Es05, Es06, Valencia
- Taiwan (5):
  - TW-02, Chiayi City
  - Tw-04, Tw-07, Kaohsiung City
  - TW-03, Taichung
  - TW-05, Tainan
  - Tw-01, Tw-06, Taipei
- United Kingdom (4):
  - GB03, Liverpool
  - GB01, Manchester
  - GB02, Milton Keynes
  - GB04, Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Acs K, Miettinen JJ, Sergeev P, Heckel T, Diao Y, Witt-Mulder K, Thureson M, Bischler T, Huppunen ME, Suvela M, Obermuller J, Munawar U, Slipicevic A, Bargou RC, Lehmann F, Gelius SS, Norin S, Schjesvold F, Sonneveld P, Stuhmer T, Heckman CA. Efficacy of melflufen in multiple myeloma with mutated or deleted TP53. Exp Hematol Oncol. 2025 Dec 23;14(1):138. doi: 10.1186/s40164-025-00729-1. PMID 41437395
- [Derived] Schjesvold FH, Ludwig H, Delimpasi S, Robak P, Coriu D, Tomczak W, Pour L, Spicka I, Dimopoulos MA, Masszi T, Chernova NG, Sandberg A, Thuresson M, Norin S, Bakker NA, Mateos MV, Richardson PG, Sonneveld P. Health-related quality of life in relapsed/refractory multiple myeloma treated with melflufen and dexamethasone: analyses from the phase III OCEAN study. Haematologica. 2024 Jul 1;109(7):2331-2336. doi: 10.3324/haematol.2023.284635. No abstract available. PMID 38426292
- [Derived] Sonneveld P, Richardson PG, Ludwig H, Dimopoulos MA, Schjesvold FH, Hajek R, Abdulhaq H, Thuresson M, Norin S, Bakker NA, Mateos MV. Benefit Versus Risk Assessment of Melflufen and Dexamethasone in Relapsed/Refractory Multiple Myeloma: Analyses From Longer Follow-up of the OCEAN and HORIZON Studies. Clin Lymphoma Myeloma Leuk. 2023 Sep;23(9):687-696. doi: 10.1016/j.clml.2023.05.004. Epub 2023 May 6. PMID 37355418
- [Derived] Schjesvold FH, Dimopoulos MA, Delimpasi S, Robak P, Coriu D, Legiec W, Pour L, Spicka I, Masszi T, Doronin V, Minarik J, Salogub G, Alekseeva Y, Lazzaro A, Maisnar V, Mikala G, Rosinol L, Liberati AM, Symeonidis A, Moody V, Thuresson M, Byrne C, Harmenberg J, Bakker NA, Hajek R, Mateos MV, Richardson PG, Sonneveld P; OCEAN (OP-103) Investigators. Melflufen or pomalidomide plus dexamethasone for patients with multiple myeloma refractory to lenalidomide (OCEAN): a randomised, head-to-head, open-label, phase 3 study. Lancet Haematol. 2022 Feb;9(2):e98-e110. doi: 10.1016/S2352-3026(21)00381-1. Epub 2022 Jan 12. PMID 35032434

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment was performed from specialized clinics' own patient pool at 115 different treatment sites in the US, Europe and Asia (20 different countries). The first patient was recruited in 12-Jun-2017 and the last patient 25-Aug-2020.
Pre-assignment Details: 246 patients were randomized to treatment Arm A, 249 patients to treatment Arm B (FAS). Of the 495 randomized patients, 228 patients in Arm A received treatment and 246 patients in Arm B received treatment (SAF). The protocol had pre-defined treatment criteria for specific laboratory values, and if the patient's values deteriorated between screening and C1D1, treatment could not be initiated. In total, 664 patients were screened, 495 randomized, 474 treated, 21 randomized but not treated.
Period: Overall Study
Arm/Group | Arm A: Melflufen+Dexamethasone | Arm B: Pomalidomide+Dexamethasone
Started | 246 | 249
Completed (Patients were to receive treatment until there was documented disease progression, unacceptable toxicity, or the patient/treating physician determined it was not in the patient's best interest to continue. The study Sponsor terminated the study before all patients reached one of these endpoints. Shown here are the reasons for study treatment discontinuation.) | 0 | 0
Not Completed | 246 | 249
Not completed — Randomized But Not Treated | 18 | 3
Not completed — Progressive Disease | 130 | 170
Not completed — Adverse Event | 49 | 40
Not completed — Lack of Efficacy | 6 | 8
Not completed — Physician Decision | 21 | 9
Not completed — Withdrawal by Subject | 17 | 7
Not completed — Lost to Follow-up | 0 | 1
Not completed — Study Terminated by Sponsor | 5 | 11

BASELINE CHARACTERISTICS:
Population: All patients that were enrolled defined as patients assigned a unique patient number by Interactive Response Technology system at the time of enrollment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Melflufen+Dexamethasone | Arm B: Pomalidomide+Dexamethasone | Total
Number analyzed (Participants) | 246 | 249 | 495
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 96 | 85 | 181
  >=65 years | 150 | 164 | 314
Age, Continuous [Median (Full Range); unit: years] | 68 [41 to 91] | 68 [39 to 87] | 68 [39 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 109 | 216
  Male | 139 | 140 | 279
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 5 | 13
  Not Hispanic or Latino | 232 | 237 | 469
  Unknown or Not Reported | 6 | 7 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 8 | 13 | 21
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 224 | 222 | 446
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 10 | 10 | 20
Region of Enrollment [Number; unit: participants]
  Romania | 10 | 10 | 20
  Hungary | 17 | 14 | 31
  Czechia | 29 | 30 | 59
  United States | 11 | 15 | 26
  United Kingdom | 5 | 5 | 10
  Spain | 22 | 20 | 42
  Russia | 40 | 39 | 79
  Greece | 23 | 23 | 46
  Netherlands | 2 | 1 | 3
  Austria | 1 | 2 | 3
  South Korea | 7 | 8 | 15
  Belgium | 3 | 2 | 5
  Norway | 14 | 19 | 33
  Taiwan | 1 | 4 | 5
  Denmark | 1 | 0 | 1
  Poland | 23 | 24 | 47
  Italy | 16 | 14 | 30
  Israel | 7 | 7 | 14
  France | 9 | 10 | 19
  Lithuania | 2 | 1 | 3
  Estonia | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Progression Free Survival defined as the duration in months from randomization until first evidence of confirmed disease progression, as assessed by the Independent Review Committee (IRC) according to the International Myeloma Working Group Uniform Response Criteria (IMWG-URC). Disease progression was defined according to the IMWG-URC as progressive disease or death due to any cause, whichever occurs first.
Time Frame: From date of randomization until first evidence of confirmed disease progression or death due to any cause (whichever occurred first), up to the data cutoff date of 03 Feb 2021 (ie, assessed up to approximately 43 months).
Population: All randomized patients (Full Analysis Set as per protocol) were included into the primary outcome measure analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Melflufen+Dexamethasone | Arm B: Pomalidomide+Dexamethasone
Number analyzed (Participants) | 246 | 249
months | 6.83 [4.96 to 8.54] | 4.93 [4.24 to 5.72]
Statistical Analysis 1: Comparison: Arm A: Melflufen+Dexamethasone vs Arm B: Pomalidomide+Dexamethasone; Test type: Superiority; p = 0.0311, Log Rank

2. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR defined as the proportion of patients for whom the best overall confirmed response is stringent complete response (sCR), complete response (CR), very good partial response (VGPR), or partial response (PR), as assessed by IRC.
Time Frame: From randomization until best response achieved before confirmed disease progression or death due to any cause, up to data cutoff of 03 Feb 2021 (ie, assessed up to approx. 43 months). Median time to best response: Arm A=2.1 months and Arm B=2.0 months
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Melflufen+Dexamethasone | Arm B: Pomalidomide+Dexamethasone
Number analyzed (Participants) | 246 | 249
Participants | 80 | 67

3. Secondary Outcome: Duration of Response (DOR)
Description: DOR defined as the duration in months from first documentation of a confirmed response to first evidence of confirmed disease progression or death due to any cause.
Time Frame: From first documentation of a confirmed response to first evidence of confirmed disease progression or death due to any cause, up to the data cutoff date of 03 Feb 2021 (ie, assessed up to approximately 43 months).
Population: Full Analysis Set (all patients randomized to either Arm A or Arm B).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Melflufen+Dexamethasone | Arm B: Pomalidomide+Dexamethasone
Number analyzed (Participants) | 246 | 249
months | 11.17 [8.48 to 17.48] | 11.07 [7.62 to 15.44]

4. Secondary Outcome: Overall Survival (OS)
Description: OS defined as the time in months from randomization to date of death due to any cause. Patients who were still alive at end of study, or lost to follow up, were censored at the last day the patient was known to be alive.
Time Frame: From date of randomization until up to 24 months following confirmed disease progression or initiation of subsequent therapy, up to the data cutoff date of 03 Feb 2023 (ie, assessed up to approximately 67 months).
Population: Full Analysis Set (all patients randomized to either Arm A or Arm B).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Melflufen+Dexamethasone | Arm B: Pomalidomide+Dexamethasone
Number analyzed (Participants) | 246 | 249
Months | 20.24 [15.84 to 24.15] | 23.98 [18.92 to 27.86]

5. Secondary Outcome: Safety and Tolerability: Number of Patients With Treatment-emergent Adverse Events (TEAEs), Including Clinical Laboratory and Vital Signs Abnormalities, as Assessed by CTCAE v4.0
Description: Number of patients with TEAEs, including clinical laboratory and vital signs abnormalities, as assessed by CTCAE v4.0 are presented. No formal statistical analysis was performed for safety endpoints.
Time Frame: From start of dosing until 30 days after the last dose of study treatment, up to the data cutoff date of 03 Feb 2023 (ie, assessed up to approximately 67 months). Median duration of study treatment was 25.2 and 22.1 weeks for Arm A and B, respectively.
Population: Safety Analysis Set (all patients that have received at least one dose of study drug in either Arm A or Arm B).
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Melflufen+Dexamethasone | Arm B: Pomalidomide+Dexamethasone
Number analyzed (Participants) | 228 | 246
Participants | 227 | 243

ADVERSE EVENTS:
Time Frame: Deaths were recorded from time of randomization until death or withdrawal from study and TEAEs were recorded from start of treatment until 30 days after the last dose of study drug, up to the data cutoff of 03 Feb 2023 (ie, assessed up to approx. 67 months). Eligibility for treatment was reconfirmed on C1D1, resulting in 18 patients never treated in Arm A and 3 patients in Arm B. Patients were treated in 28-day cycles indefinitely until withdrawal from study. Longest time on study was 60 months.
Description: All-cause mortality is reported for the Full Analysis Set (all randomized patients; Arm A=246 patients, Arm B=249 patients). Adverse Events are reported for the Safety Analysis Set (all patients who received at least one or partial dose of melflufen, pomalidomide, or dexamethasone; Arm A=228 patients, Arm B=246 patients). Non-serious AEs were not calculated in this study. Data reported in the "Other Adverse Events" section include all TEAEs (non-serious AEs and serious AEs).
Arm/Group | Arm A: Melflufen+Dexamethasone | Arm B: Pomalidomide+Dexamethasone
All-Cause Mortality (participants affected / at risk) | 180/246 | 169/249
Serious Adverse Events (participants affected / at risk) | 99/228 | 124/246
Other Adverse Events (participants affected / at risk) | 227/228 | 243/246
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Melflufen+Dexamethasone (N=228) | Arm B: Pomalidomide+Dexamethasone (N=246)
Pneumonia (Infections and infestations) | 14 (17) | 23 (26)
COVID-19 pneumonia (Infections and infestations) | 12 (13) | 14 (14)
Urinary tract infection (Infections and infestations) | 2 (2) | 6 (11)
Sepsis (Infections and infestations) | 1 (1) | 6 (6)
Bronchitis (Infections and infestations) | 3 (4) | 4 (5)
Influenzae (Infections and infestations) | 0 (0) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 1 (1)
Viral Infection (Infections and infestations) | 1 (3) | 3 (3)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 3 (4)
Respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2)
Septic shock (Infections and infestations) | 0 (0) | 3 (3)
Escherichia sepsis (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Infection (Infections and infestations) | 2 (2) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 1 (1)
Abscess jaw (Infections and infestations) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Arthritis fungal (Infections and infestations) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Bacterial sepsis (Infections and infestations) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Lymphangitis (Infections and infestations) | 1 (1) | 0 (0)
Moraxella infection (Infections and infestations) | 1 (1) | 0 (0)
Muscle abscess (Infections and infestations) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0)
Orchitis (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Parainfluenzae virus infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 1 (3)
Pneumonia streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 8 (11) | 6 (13)
Thrombocytopenia (Blood and lymphatic system disorders) | 11 (15) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 5 (6) | 3 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (5) | 2 (2)
Pancytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
General physical health deterioration (General disorders) | 2 (2) | 4 (5)
Pyrexia (General disorders) | 5 (6) | 3 (3)
Multiple organ dysfunction syndrome (General disorders) | 2 (2) | 2 (2)
Asthenia (General disorders) | 1 (1) | 1 (2)
Chest Pain (General disorders) | 1 (1) | 1 (1)
Pain (General disorders) | 1 (1) | 1 (1)
Sudden cardiac death (General disorders) | 0 (0) | 2 (2)
Administration site extravasion (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Sudden death (General disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4)
Pumlonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 3 (3)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 9 (11)
Cardiac arrest (Cardiac disorders) | 2 (2) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Cardiovascular insufficiency (Cardiac disorders) | 0 (0) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Sternal fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Oesophageal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Abdominal mass (Gastrointestinal disorders) | 2 (2) | 0 (0)
Cholitis ischaemic (Gastrointestinal disorders) | 1 (2) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Obstructive pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oral mucosal hypertrophy (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis chronic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (3)
Renal Failure (Renal and urinary disorders) | 2 (2) | 6 (6)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 5 (5)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (4)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Vertebral lesion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 3 (3)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 1 (1)
Brain oedema (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular insufficiency (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 1 (1)
Monoplegia (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 4 (5) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (3)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 2 (2)
Circulatory collapse (Vascular disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Thrombophlebitis superficial (Vascular disorders) | 1 (1) | 0 (0)
Hypercalcaemia of malignancy (Endocrine disorders) | 1 (1) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 3 (3)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 1 (2)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Device related sepsis (Infections and infestations) | 1 (1) | 0 (0)
Rhinovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pathological fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cerebral venous sinus thrombosis (Nervous system disorders) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Post stroke epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Vascular encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Panniculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Melflufen+Dexamethasone (N=228) | Arm B: Pomalidomide+Dexamethasone (N=246)
Neutropenia (Blood and lymphatic system disorders) | 137 (795) | 115 (421)
Anaemia (Blood and lymphatic system disorders) | 154 (487) | 97 (238)
Thrombocytopenia (Blood and lymphatic system disorders) | 161 (918) | 50 (149)
Leukopenia (Blood and lymphatic system disorders) | 24 (89) | 11 (18)
Diarrhoea (Gastrointestinal disorders) | 32 (46) | 24 (32)
Nausea (Gastrointestinal disorders) | 31 (44) | 18 (20)
Constipation (Gastrointestinal disorders) | 17 (19) | 29 (33)
Fatigue (General disorders) | 33 (52) | 44 (57)
Asthenia (General disorders) | 33 (50) | 32 (47)
Pyrexia (General disorders) | 33 (43) | 18 (25)
Oedema peripheral (General disorders) | 12 (17) | 24 (24)
Upper respiratory tract infection (Infections and infestations) | 29 (33) | 27 (43)
Bronchitis (Infections and infestations) | 13 (16) | 29 (42)
Pneumonia (Infections and infestations) | 21 (26) | 36 (47)
Urinary tract infection (Infections and infestations) | 12 (17) | 16 (24)
Respiratory tract infection (Infections and infestations) | 8 (12) | 20 (24)
COVID-19 pneumonia (Infections and infestations) | 12 (15) | 14 (16)
Neutrophil count decreased (Investigations) | 30 (154) | 28 (88)
Platelet count decreased (Investigations) | 40 (198) | 11 (25)
White blood cell count decreased (Investigations) | 22 (86) | 6 (9)
SARS-CoV-2 test positive (Investigations) | 16 (17) | 22 (26)
Back pain (Musculoskeletal and connective tissue disorders) | 19 (20) | 26 (33)
Bone pain (Musculoskeletal and connective tissue disorders) | 16 (18) | 13 (19)
Athralgia (Musculoskeletal and connective tissue disorders) | 16 (20) | 8 (9)
Dizziness (Nervous system disorders) | 8 (9) | 16 (21)
Insomnia (Psychiatric disorders) | 21 (23) | 21 (29)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 22 (27) | 27 (28)
Cough (Respiratory, thoracic and mediastinal disorders) | 20 (24) | 20 (30)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 14 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-04-20): https://cdn.clinicaltrials.gov/large-docs/11/NCT03151811/Prot_002.pdf
  • Statistical Analysis Plan (2021-10-25): https://cdn.clinicaltrials.gov/large-docs/11/NCT03151811/SAP_003.pdf